CLINICAL TRIAL: NCT02478827
Title: A Trial of Cognitive Training in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Vina M. Goghari, Dr. Vina Goghari, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: REB15-0526
Record Dates: First submitted 2015-06-15; First posted 2015-06-23 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
Keywords: Cognitive Training; Working Memory; Processing Speed
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Working Memory group (Experimental): The neurocognitive training program will be provided by an online platform called BrainGymmer (https://www.braingymmer.com/en/brain-games/). Users will receive an account where they will only have access to the training games they have been assigned to and where their activity will be logged. One experimental group will complete the working memory training, which involves three games: N-back, Multi-Memory, and Moving Memory. These games are designed to engage processes involving updating and manipulation of information. All of the training games are adaptive. Participants randomized to this cognitive training arm will complete the training games for 30 minutes per day, 5 days a week, for a total of 10 weeks.
  Interventions: Behavioral: Cognitive training
- Processing Speed group (Experimental): The neurocognitive training program will be provided by an online platform called BrainGymmer (https://www.braingymmer.com/en/brain-games/). Users will receive an account where they will only have access to the training games they have been assigned to and where their activity will be logged. One experimental group will complete the processing speed training, which involves three games: Line It Up, Sliding Search, and Bubble Math. These games are designed to engage processes involving thinking speed. Participants randomized to this cognitive training arm will complete the training games for 30 minutes per day, 5 days a week, for a total of 10 weeks
  Interventions: Behavioral: Cognitive training
- Control group (No Intervention): The control group will wait 10-weeks, during which they will receive treatment-as-usual (TAU), which might involve pharmacotherapy, psychotherapy, or both. After the 10-week waiting period, a post-assessment will be completed.

INTERVENTIONS:
Behavioral: Cognitive training — The neurocognitive training program will be provided by an online platform called BrainGymmer (https://www.braingymmer.com/en/brain-games/). Users will receive an account where they will only have access to the training games they have been assigned to and where their activity will be logged. Participants randomized one of the cognitive training arms will complete the training games for 30 minutes per day, 5 days a week, for a total of 10 weeks.
  Arms: Processing Speed group; Working Memory group

SUMMARY:
Schizophrenia is associated with a wide range of symptoms impacting a number of different domains, including cognitive impairment. Given the array of cognitive deficits associated with schizophrenia and their relationship to daily functioning, numerous research groups have examined the impact of cognitive remediation on many aspects of cognition. However, it is currently unclear as to which domains of cognition should be targeted to produce the most widespread and durable benefits for schizophrenia patients. It may be the case that targeting lower-level cognitive processes that are important for higher-level and more complex aspects of cognition may produce the most widespread benefits in cognition and everyday functioning. Relatively few studies have examined the effects of working memory or processing speed training on individuals with schizophrenia, as most studies examine broad-based remediation programs. Thus, there is a need for targeted working memory and processing speed training studies to better understand the mechanisms of cognitive enhancement through training in patients. This study will aim to: 1) investigate near-transfer gains associated with working memory and processing speed training in schizophrenia patients, 2) investigate far-transfer gains associated with working memory and processing speed training (i.e., gains in other neurocognitive domains and social cognition), and 3) investigate real-world gains associated with training (i.e., gains in daily functioning). Towards this aim, 81 schizophrenia patients will be recruited and randomly assigned to a working memory training group, a processing speed training group, or a no training control group. Training will be completed at home for 30 minutes per day, 5 days per week, for a total of 10 weeks. Neurocognitive, social cognitive, and daily functioning measures will be administered both pre- and post-training to detect training-related gains.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age between 18 and 65 years
* A diagnosis of schizophrenia or schizoaffective disorder
* Minimum IQ of 70
* No uncorrected visual impairment, including colour blindness
* No uncorrected hearing impairment
* Able to provide informed consent

Exclusion Criteria:

* Meeting Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) diagnostic criteria for a current major depressive episode, manic episode, or hypomanic episode
* Past 1 month history of electroconvulsive therapy (ECT)
* Past 1 month history of Transcranial Magnetic Stimulation therapy (TMS)
* Past 3 month history of substance abuse
* Diagnosed with a medical condition known to affect cognition (e.g., endocrine disease)
* Score less than 70 on the Wechsler Abbreviated Scale of Intelligence (WASI)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Fluid intelligence | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with Raven's Standard Progressive Matrices and Cattell's Culture Fair Test
Working Memory | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with Wechsler Adult Intelligence Scale 4th Edition (WAIS-IV) Digit Span, Spatial Maintenance and Manipulation Task, and Visual N-Back Task
Processing Speed | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with Wechsler Adult Intelligence Scale 4th Edition (WAIS-IV) Symbol Search and Delis-Kaplan Executive Function System (D-KEFS) Color Naming Task

SECONDARY OUTCOMES:
Executive functions: categorization, set-shifting, and cognitive flexibility | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with Delis-Kaplan Executive Function System (D-KEFS) Color-Word Interference Test and Trail Making Test
Behavioural Impulsivity | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with Delay Discounting Task

OTHER OUTCOMES:
Social Cognition: Emotion Recognition and Theory of Mind | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with Geneva Emotion Recognition Test and Hinting Task
Daily functioning: cognitive failures in daily life, performance, social, and occupational functioning | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with Cognitive Failures Questionnaire, UCSD Performance-Based Skills Assessment (UPSA-Brief), and Social and Occupational Functional Assessment Scale (SOFAS)
Symptoms | Change from baseline to post-assessment (after 10 weeks of training)
  Measured with Positive and Negative Syndrome Scale (PANSS)
Beliefs Regarding Cognition | Change from baseline to post-assessment (after 10 weeks of training)
  Need for Cognition Scale and Theories of Intelligence Scale

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Foothills Medical Centre, Calgary, Alberta
  - Schizophrenia Society of Alberta, Calgary
  - Schizophrenia Society of Alberta, Edmonton

REFERENCES:
- [Background] Lawlor-Savage L, Goghari VM. Working memory training in schizophrenia and healthy populations. Behav Sci (Basel). 2014 Sep 3;4(3):301-319. doi: 10.3390/bs4030301. eCollection 2014 Sep. PMID 25379283
- [Derived] Cassetta BD, Goghari VM. Working memory and processing speed training in schizophrenia: study protocol for a randomized controlled trial. Trials. 2016 Jan 26;17:49. doi: 10.1186/s13063-016-1188-5. PMID 26812902